CLINICAL TRIAL: NCT03423108
Title: Exercise Dose-response for Diabetes in the Elderly: a Randomized Clinical Trial.
Brief Title: Exercise Dose-response for Diabetes in the Elderly
Acronym: EDDIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0303
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-03

CONDITIONS: Type2 Diabetes
Keywords: Exercise; Aging; Elderly; Physical Activity; Cardiovascular Disease
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants randomized to this group will perform monthly cohabitation meetings.
- G150 (Experimental): Participants randomized to this group will be enrolled to a 150 min/week structured and supervised exercise training. The program consists of 3 sessions in a week, each of these lasting 50 minutes. The session will be composed of aerobic training (25 minutes at 60-75% of HRmax) and strength training (25 minutes, 8 whole-body exercises at up to 8-12 maximal repetitions).
  Interventions: Behavioral: G150
- G300 (Experimental): Participants randomized to this group will be enrolled to the same structural settings of G150 group (type of exercise, exercise intensity and weekly frequency). They will receive twice the G150 group dose's. To do so, each session will last 100 minutes (50 minutes of aerobic exercise training and 50 minutes of strength training).
  Interventions: Behavioral: G300

INTERVENTIONS:
Behavioral: G150 — This group will receive 150 min/week of combined exercise training, structured and supervised.
  Arms: G150
Behavioral: G300 — This group will receive 300 min/week of combined exercise training, structured and supervised.
  Arms: G300

SUMMARY:
One-center randomized, three-arm, parallel, superiority, controlled trial in 132 elderly outpatients with type 2 diabetes. Two different combined exercise training doses (300min/week vs 150min/week) will be compared against usual care. The entire study length will last 24 weeks, and assessments will be conducted at baseline, previously to the group allocation, at 12 weeks and at 24 weeks just after the treatments' end. The study's primary outcome is the glycated hemoglobin level at 24 weeks. Secondary outcomes of clinical relevance to type 2 diabetes and elderlies will also be acquired.

DETAILED DESCRIPTION:
This study is a randomized controlled trial, three-arm parallel-group. The first aim is to evaluate the efficacy of a supervised and structured combined exercise training program in HbA1c levels at 24 weeks. Secondary outcomes measurements of clinical relevance for type 2 diabetes and elderly patients are included at 12 and 24 weeks.

The investigators will enroll 132 elderlies divided into three experimental groups, randomized in a ratio of 1:1 (44 patients per group). The treatments arms comprises structured supervised combined exercise training programs, three times a week, lasting 24 weeks of duration. The G150 group will exercise 150 min per week of aerobic and strength training (50 min per session, 25 min for each modality) and the G300 group will exercise twice the volume in the same G150's intensity, and week frequency (100 min per session, 50 min for each modality). No intervention will be offered to the control group (i.e., they will continue their usual care). Treatments arms will progress on training load tailored by their maximal heart rate percentage for aerobic training and maximal repetitions for strength training.

The sample size was calculated considering a between-group mean difference of 0.45%, with standard deviation of 0.7% in HbA1c levels, for an 80% of statistical power and 5% of type 1 error, in a superiority hypothesis design.

In detail, the primary outcome is the HbA1c level at 24 weeks, an secondary outcomes are: HbA1c levels at 12 weeks; office blood pressure assessed through a digital sphygmomanometer at 12 and 24 weeks; lipid profile (total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides) at 24 weeks; endothelial function assessed by flow-mediated dilation at 12 and 24 weeks; intima-media thickness at 24 weeks; physical fitness assessed by maximal oxygen uptake and maximal muscle strength at 24 weeks; body composition assessed by dual x ray absorptiometry at 24 weeks; quality of life and geriatric depressive symptoms assessed by questionnaires at 24 weeks.

The investigators hypothesized that the G300 will greater improve the 24-week HbA1c levels and secondary outcomes against the G150 and the control group. The present study was designed and will be conducted by a multidisciplinary staff, and follows ethical and methodological standards for randomized clinical trials. As for empirical evidence provision, it is expected to highlight the efficacy of the non-pharmacological treatment for type 2 diabetes in the elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of type 2 diabetes mellitus by HbA1c (> 6.5%) or capillary casual glycemia (> 126 mg/dL), oral glucose tolerance test or hypoglycemic drug use;
* HbA1c ≥ 7.5%;
* Verified ability to exercise;
* Physically inactive or regularly exercising for at least once a week.

Exclusion Criteria:

* HbA1c ≤ 12%;
* Severe cardiovascular disease (class III or IV heart failure, uncontrolled arrhythmia, unstable angina, or use of implantable cardioverter defibrillator);
* Major cardiovascular events 1 year previously to the enrollment (non-fatal myocardial infarction, coronary artery bypass surgery, cardiac catheterization, deep vein thrombosis, hospitalization or other severe health-related event);
* Chronic renal disease requesting dialysis;
* Severe macular injury (retinopathy) that disables patients to enroll an exercise program;
* Severe cognitive impairment (dementia) that disables patients to enroll an exercise program;
* Deafness that disables patients to enroll an exercise program;
* Blindness that disables patients to enroll an exercise program;
* Progressive neurological disorders (Parkinson, multiple sclerosis, etc.) that disables patients to enroll an exercise program;
* Osteoarticular or muscular injuries or another health conditions which generate inability to carry on the interventions;
* Plans of moving to another city during the study;
* Living together with another person enrolled in the study;
* A medical report indicating exercise contraindication based on a cardiopulmonary exercise testing;
* Inability or refusal to give written consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2018-09-10 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Change from baseline to 24 weeks
  Glycated hemoglobin in DCCT units (%)

SECONDARY OUTCOMES:
HbA1c | Change from baseline to 12 weeks
  Glycated hemoglobin in DCCT units (%)
Office Blood Pressure | Change from baseline to 12 weeks
  Systolic and diastolic blood pressure measured through automatic oscillometric device in mmHg
Office Blood Pressure | Change from baseline to 24 weeks
  Systolic and diastolic blood pressure measured through automatic oscillometric device in mmHg
Lower limbs functional capacity | Change from baseline to 24 weeks
  By using the Short Physical Performance Battery (SPPB), lower-limb mobility will be assess in the following sequence: static standing balance, walking speed and indirect muscle strength. The performance of functional activities will be converted to a standardized scale from 0 (poor functional capacity) to 12 points (excellent functional capacity)
Cardiorespiratory fitness | Change from baseline to 24 weeks
  Peak oxygen uptake (VO2peak) assessed by maximal cardiopulmonary exercise testing and reported in its weighted form (ml/kg/min)
Geriatric Depression Symptoms | Change from baseline to 24 weeks
  Geriatric depression alertness and improvements will be assessed through a questionnaire comprised by 15 questions in a YES/NO answer options nested to 0/1 numbered options. Alertness of geriatric depression is characterized when the overall score reaches 5 points or below it. The overall score is calculated a posteriori due to variations on questions directions (e.g., YES = 1 or YES = 0 conditioned to the question).
Endothelial function, early adaptation | Change from baseline to 12 weeks
  Flow-mediated dilatation (FMD) assessed through high resolution ultrasonography
Endothelial function | Change from baseline to 24 weeks
  Flow-mediated dilatation (FMD) assessed through high resolution ultrasonography
Intima-media thickness | Change from baseline to 24 weeks
  Intima-media thickness (IMT) assessed through high resolution ultrasonography
Body composition | Change from baseline to 24 weeks
  Body composition assessed by dual x-ray absorptiometry system (DXA)
Quality of life (QoL) | Change from baseline to 24 weeks
  Patients' quality of life will be assessed by the World Health Organization Quality of Life for Elderlies (WHOQoL-OLD) instrument. It comprises 24 questions and answers are presented in a one-way direction, 1-to-5 scale.
Muscle thickness | Change from baseline to 24 weeks
  Muscle thickness assessed through high resolution ultrasonography
Muscle quality | Change from baseline to 24 weeks
  Image echo-intensity assessed through high resolution ultrasonography
Lower body maximal muscle strength | Change from baseline to 24 weeks
  Lower body maximal muscle strength will be assessed by the knee extension one-maximal repetition test, reported in kilograms (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Umpierre, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre/Federal University of Rio Grande do Sul; Beatriz Schaan, MD, PhD, Study Director — Hospital de Clinicas de Porto Alegre/Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data HbA1c and neuromuscular function and any deemed relevant support information (sociodemographic, clinical history and allocated groups) will be shared if available. Details regarding the study's design and statistical plan can be obtained consulting the trial's protocol. Data on other outcomes could be requested contacting the PI. Data access will be available after all participants completed the study and will remain accessible for as long as deemed necessary by the study's committee. Data sets, variables' dictionary and statistical analysis description will be made available online upon registration at a clinical trial management system nested to the EDDIE Study's website (www.ufrgs.br/eddie), and the access will be permitted after acceptance of the EDDIE Study team's data sharing terms and policy.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The individual participant dataset will become available up to six months after the first study publication.
Access Criteria: A simple registration aside a policy acceptance term will grant access to study's datasets.
URL: http://www.ufrgs.br/eddie